CLINICAL TRIAL: NCT02975739
Title: Feasibility of Holmium-166 Microspheres for Selective Intra-tumoural Treatment in Head and Neck Cancer: Biodistribution and Safety in Patients With Malignancy of the Tongue
Brief Title: Feasibility of Holmium-166 Micro Brachytherapy in Head and Neck Tumors
Acronym: HIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Marnix Lam, Professor Nuclear medicine, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL54535.041.15
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Radioisotopes; Head and Neck Neoplasms
Keywords: Intratumoral; Tongue; Microspheres
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Microspheres

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Holmium-166 microspheres (Experimental): Single session of 4 intratumoral injections consisting of 0.1-0.3 ml radioactive Holmium-166 microsphere suspension with a total activity 30 Megabecquerel, 7-12 days prior to surgical resection.
  Interventions: Device: Holmium-166 (poly L lactic acid) microspheres

INTERVENTIONS:
Device: Holmium-166 (poly L lactic acid) microspheres — Intratumoral injections of Holmium-166 (poly L lactic acid) microspheres
  Other Names: Holmium microspheres

SUMMARY:
The main objective is to establish the feasibility of 166-Holmium microspheres for intratumoral injections in oral squamous cell carcinoma (OSCC) of the tongue.

Participants will receive intratumoral injections with a low radioactive 166-Holmium microspheres followed by surgical resection

DETAILED DESCRIPTION:
166-Holmium microspheres poly lactic acid microspheres are currently used in selective internal radiation therapy. These microspheres emits beta radiation. The majority of the radiation dose will be absorbed within 3.2 mm with a maximum penetration in tissue of 9 mm. Therefore this can result in a high local tumor ablative dose with minimal dose to healthy adjacent tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have given written informed consent.
2. Aged 18 years and over.
3. Confirmed histological diagnosis of squamous cell carcinoma of the tongue.
4. primary tumor, regional nodes, metastasis (TNM) stage T1-2 Nx M0.
5. Eligible for local surgery with curative intent.
6. World Health Organization (WHO) Performance status 0-2.

Exclusion Criteria:

1. Previous oncologic surgery and/or external beam radiation therapy on the tongue and oral floor.
2. Major surgery (Oro-facial) within the past 4 weeks or incompletely healed surgical incisions before starting study therapy.
3. Any unresolved toxicity greater than National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE version 4.03) grade 2 from previous anti-cancer therapy.
4. Pregnancy or nursing (women of child-bearing potential).
5. Patients suffering from psychic disorders that make a comprehensive judgment impossible, such as psychosis, hallucinations and/or depression.
6. Previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Total amount of activity leakage (in percentage) in the oral cavity rinsing fluid. | upto 5 minutes after administration

SECONDARY OUTCOMES:
Occurrence of (serious) adverse events | Between administration and resection of the tumor (max 12 days)
The biodistribution of Holmium-166 microspheres after intra-tumoural injection | upto 30 minutes after administration
  SPECT Thorax and Abdomen Radioactivity in a blood and urine sample
The biodistribution of Holmium-166 microspheres after intra-tumoural injection | 1-2 hours after administration
  MRI
The biodistribution of Holmium-166 microspheres after intra-tumoural injection | 3 hours after administration
  Radioactivity in blood and urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Marnix G Lam, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Es RJ, Nijsen JF, van het Schip AD, Dullens HF, Slootweg PJ, Koole R. Intra-arterial embolization of head-and-neck cancer with radioactive holmium-166 poly(L-lactic acid) microspheres: an experimental study in rabbits. Int J Oral Maxillofac Surg. 2001 Oct;30(5):407-13. doi: 10.1054/ijom.2001.0129. PMID 11720043
- [Background] Bult W, Vente MA, Vandermeulen E, Gielen I, Seevinck PR, Saunders J, van Het Schip AD, Bakker CJ, Krijger GC, Peremans K, Nijsen JF. Microbrachytherapy using holmium-166 acetylacetonate microspheres: a pilot study in a spontaneous cancer animal model. Brachytherapy. 2013 Mar-Apr;12(2):171-7. doi: 10.1016/j.brachy.2012.08.001. Epub 2012 Sep 19. PMID 22999975
- [Background] Smits ML, Nijsen JF, van den Bosch MA, Lam MG, Vente MA, Mali WP, van Het Schip AD, Zonnenberg BA. Holmium-166 radioembolisation in patients with unresectable, chemorefractory liver metastases (HEPAR trial): a phase 1, dose-escalation study. Lancet Oncol. 2012 Oct;13(10):1025-34. doi: 10.1016/S1470-2045(12)70334-0. Epub 2012 Aug 22. PMID 22920685
- [Background] Bult W, de Leeuw H, Steinebach OM, van der Bom MJ, Wolterbeek HT, Heeren RM, Bakker CJ, van Het Schip AD, Hennink WE, Nijsen JF. Radioactive holmium acetylacetonate microspheres for interstitial microbrachytherapy: an in vitro and in vivo stability study. Pharm Res. 2012 Mar;29(3):827-36. doi: 10.1007/s11095-011-0610-7. Epub 2011 Nov 9. PMID 22068276